CLINICAL TRIAL: NCT04365101
Title: A Phase I/II Study of Human Placental Hematopoietic Stem Cell Derived Natural Killer Cells (CYNK-001) for the Treatment of Adults With COVID-19
Brief Title: Natural Killer Cell (CYNK-001) Infusions in Adults With COVID-19
Acronym: CYNKCOVID
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Celularity Incorporated (Industry)
Collaborators: Access to Advanced Health Institute (AAHI) (Other); Lung Biotechnology PBC (Industry); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYNK-001-COVID-19
Record Dates: First submitted 2020-04-22; First posted 2020-04-28 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Coronavirus; Coronavirus Infection; Severe Acute Respiratory Syndrome Coronavirus 2; Pneumonia; Pneumonia, Viral; Lung Diseases; Respiratory Tract Disease; Respiratory Tract Infections; Coronaviridae Infections; Nidovirales Infections; RNA Virus Infections; Virus Disease; Immunologic Disease; ARDS; Immunologic Factors; Physiological Effects of Drugs; Antiviral Agents; Anti-infective Agents; Analgesics; Antimetabolites, Antineoplastic
Keywords: CYNK-001; Coronavirus; COVID-19; SARS-Cov-2; cell therapy; NK cells; natural killer cells; CYNKCOVID; CYNK-001-COVID-19
MeSH Terms: conditions — Coronavirus Infections; Pneumonia; Pneumonia, Viral; Lung Diseases; Respiratory Tract Diseases; Respiratory Tract Infections; Coronaviridae Infections; Nidovirales Infections; RNA Virus Infections; Virus Diseases; Immune System Diseases; COVID-19

STUDY DESIGN:
Intervention Model Description: Phase I will evaluate the safety and efficacy of multiple doses of CYNK-001 (Days 1,4, and 7) in 14 patients.
  Phase II will utilize a randomized, open-label design; multiple doses of CYNK-001 will be compared to the control group: Best Supportive Care. Up to 72 patients will be included in the Phase II portion of the study with a 1:1 randomization ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I (Experimental): CYNK-001 infusions on Days 1, 4, and 7
  Interventions: Biological: CYNK-001
- Phase II (Active Comparator): Randomized, open label; CYNK-001 infusions on Days 1, 4, and 7 compared to Control Group: Best Supportive Care
  Interventions: Biological: CYNK-001

INTERVENTIONS:
Biological: CYNK-001 — CYNK-001 is an allogeneic off the shelf cell therapy enriched for CD56+/CD3- NK cells expanded from human placental CD34+ cells.

SUMMARY:
This study is a Phase 1 / 2 trial to determine the safety and efficacy of CYNK-001, an immunotherapy containing Natural Killer (NK) cells derived from human placental CD34+ cells and culture-expanded, in patients with moderate COVID-19 disease.

ELIGIBILITY:
Patient Inclusion Criteria:

* Patient has confirmed positivity for SARS-CoV-2 as measured by rRT-PCR or other approved test to detect SAR-CoV-2 per institutional practice.
* Patient is experiencing any symptom/clinical sign of COVID-19 illness or has a positive disease-related chest x-ray/CT scan at screening.
* Patient is ≥ 18 years of age at the time of signing the Study informed consent form (ICF).
* Patient understands and voluntarily signs the Study ICF prior to any study-related assessments/procedures are conducted.
* Patient is willing and able to adhere to the study schedule and other protocol requirements.
* SpO2 ≥ 88% on room air; oxygen is permitted as delivered by nasal cannula and/or face mask at any flow rate to achieve this SpO2. Patients must have an SpO2 ≥ 92% if on supplementary oxygen.
* Ability to be off immunosuppressive drugs for 3 days prior to infusion, unless clinically indicated. Steroids are permitted if clinically indicated and at the discretion of the treating physician. If clinically indicated, careful consideration should be taken regarding the timing and tapering of high-dose steroids.
* Female of childbearing potential (FCBP)* must not be pregnant and agree to not becoming pregnant for at least 28 days following the last infusion of CYNK-001. FCBP must agree to use an adequate method of contraception during the treatment period.

  * FCBP is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Male Patients must agree to use a condom during sexual contact for at least 28 days following the last infusion of CYNK-001, even if he has undergone a successful vasectomy.

Patient Exclusion Criteria

* Patient requires supplemental oxygen delivered by mechanical ventilation, either invasive or bilevel positive airway pressure.
* Patient admitted to Intensive Care Unit / Pulmonary Acute Care Unit designated area with severe pulmonary pneumonia, ARDS or Sepsis.
* Patient is pregnant or breastfeeding.
* Patient has a history of chronic asthma requiring ongoing medical therapy or other chronic pulmonary disease that, at the discretion of the treating physician, would contraindicate participation in this study.
* Patient has any other organ dysfunction [Common Terminology Criteria for AEs (CTCAE) Version 5.0 Grade 3] that will interfere with the administration of the therapy according to this protocol.
* Patient has inadequate organ function as defined below at time of Treatment Eligibility Period:

  1. Patient has aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase ≥ 5 x the upper limit of normal (ULN). (It is anticipated that the infection may impact liver.)
  2. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m^2 as calculated using the Modification of Diet in Renal Disease Study equation (Levey, 2006) or history of an abnormal eGFR < 60. A decline of > 15 mL/min/1.73 m^2 below normal in the past year prior to infection. (It is anticipated that the infection may impact renal function.)
  3. Patient has a bilirubin level > 2 mg/dL (unless Patient has known Gilbert's Syndrome).
* Patient has a known sensitivity or allergy to treatment additives or diluent substances of dimethyl sulfoxide (DMSO), PlasmaLyte A or human serum albumin (HSA). Please refer to investigational brochure (IB).
* Patient has active autoimmune disease other than controlled connective tissue disorder or those who are not on active therapy.
* Patient is immunocompromised, has known human immunodeficiency virus (HIV) positivity, or has actively been treated with immunosuppressive products prior to being infected with SARS-CoV-2.
* Patient has known active malignancy, unless the Patient has been free of disease for > 3 years from the date of signing the ICF. Exceptions include the following noninvasive malignancies:

  1. Basal cell carcinoma of the skin
  2. Squamous cell carcinoma of the skin
  3. Carcinoma in situ of the cervix
  4. Carcinoma in situ of the breast
  5. Incidental histological finding of prostate cancer (TNM stage of T1a or T1b)
* Detection of other respiratory viruses from mucosal surfaces that would interfere with the study treatment plan; detection of another respiratory virus is not in itself an exclusion criteria unless the investigator believes it would interfere with administration of CYNK-001.
* Patient must not have a history of unconsciousness or hemoptysis within 2 weeks of signing informed consent form.
* Patients must not have a history of unconsciousness or hemoptysis within 2 weeks of signing ICF.
* Patients must not have end stage liver disease and/or cirrhosis.
* Patient has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from participating in the study.
* Patient has any condition including the presence of laboratory abnormalities which places the patient at unacceptable risk if he or she were to participate in the study.
* Patient has any condition that confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Frequency and Severity of Adverse Events (AE) | Up to 6 months
  Number and severity of adverse events
Phase 1 Futility Check for go/no decision to move to Phase 2: Rate of clinical improvement | Study Day 15
  Proportion of patients who improved clinical symptoms as measured by the Ordinal Scale for Clinical Improvement (OSCI)
Phase 2: Time to Clinical Improvement by Ordinal Scale for Clinical Improvement (OSCI) | Study Day 28
  Time to clinical improvement measured by OSCI

SECONDARY OUTCOMES:
Rate of Clearance of SARS-CoV-2 | Study Day 28
  Proportion of patients with "negative" measurement of COVID-19 by rRT-PCR
Time to Clearance of SARS-CoV-2 | Study Day 28
  Time to clearance of SARS-CoV-2 by rRT-PCR testing of mucousal samples with "negative" measurement of COVID-19 by rRT-PCR
Phase 2: Frequency and Severity of Adverse Events (AE) | up to 6 months
  Number and severity of adverse events
Overall Clinical Benefit by time to medical discharge | up to 6 months
  Time to medical discharge as an assessment of overall clinical benefit
Overall Clinical Benefit by hospital utilization | up to 6 months
  Hospital utilization will be measured as an assessment of overall clinical benefit
Overall Clinical Benefit by measuring mortality rate | up to 6 months
  Mortality rate will be measured as an assessment of overall clinical benefit
Impact of CYNK-001 on sequential organ failure assessment (SOFA) score | Up to 28 days
  Assess the impact of CYNK-001 on changes in sequential organ failure assessment (SOFA) score.
Time to Pulmonary Clearance | Up to 28 days
  Time from randomization to the date of disappearance of virus from lower respiratory tract infection (LRTI) specimen where it has previously been found (induced sputum, endotracheal aspirate).
Rate of Pulmonary Clearance | Up to 28 days
  Proportion of patients who had disappearance of virus from lower respiratory tract infection (LRTI) specimen where it has previously been found.
Supplemental oxygen-free days | Up to 28 days
  For ventilatory support patients, the days with supplemental oxygen-free.
Proportion of patients requiring ventilation | Up to 28 days
  Proportion of patients who need invasive or non-invasive ventilation
Duration of hospitalization | Study Day 28
  Time from hospitalization to medical discharge
Radiologic Evaluation Score | Study Day 28 and Month 6
  Chest x-ray and/or CT scan results will be evaluated and scored
All-cause mortality rate | Study Day 28 and Month 6
  Proportion of patients who died
Time to clinical improvement by NEWS2 Score | Study Day 28
  Time to clinical improvement measured by NEWS2 Score
Rate of clinical improvement by NEWS2 Score | Study Day 28
  Proportion of patients who achieved clinical symptom improvement measured by NEWS2 Score

CONTACTS AND LOCATIONS:
Overall Officials: Corey Casper, MD MPH, Principal Investigator — Access to Advanced Health Institute (AAHI)
Locations (7):
- United States (7):
  - UC Irvine, Irvine, California
  - UC Davis Medical Center, Sacramento, California
  - Scripps Health, San Diego, California
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Atlantic Health, Morristown, New Jersey
  - Atlantic Health, Summit, New Jersey
  - Multicare Health System, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, Kusek JW, Van Lente F; Chronic Kidney Disease Epidemiology Collaboration. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006 Aug 15;145(4):247-54. doi: 10.7326/0003-4819-145-4-200608150-00004. PMID 16908915